CLINICAL TRIAL: NCT00248183
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter Study To Evaluate The Efficacy, Safety, And Tolerability Of PRX-00023 In Patients With Generalized Anxiety Disorder (GAD)
Brief Title: A Study To Evaluate PRX-00023 In Patients With Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Epix Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRX-CP-007
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — naluzotan

INTERVENTIONS:
Drug: PRX-00023

SUMMARY:
This is a randomized, double-blind, placebo controlled, multi-center outpatient study, in adults with GAD.

Patients 18-65 years of age, with the diagnosis of GAD according to DSM-IV criteria, who fulfill the inclusion/exclusion criteria, will be enrolled in this study.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, multi-center outpatient study, in adults with GAD.

Patients 18-65 years of age, with the diagnosis of GAD according to DSM-IV criteria, who fulfill the inclusion/exclusion criteria, will be enrolled in this study.

This is a randomized, double-blind, placebo controlled, multi-center outpatient study, in adults with GAD.

Patients 18-65 years of age, with the diagnosis of GAD according to DSM-IV criteria, who fulfill the inclusion/exclusion criteria, will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, 18-65 years of age
* Meet DSM-IV diagnostic criteria for Generalized Anxiety Disorder (GAD)
* Have a total score of ≥ 20 on the HAM-A and a score of ≥ 2 on Items 1 and 2 (anxious mood and tension) of the HAM-A
* Have no more than a 20% decrease in total HAM-A score during the period from the screening visit to the randomization visit
* Have a negative serum (β-HCG) pregnancy test at screening and a negative urine pregnancy test at baseline (for all women)
* Female subjects must meet one of the following criteria: (a) Be surgically sterile (i.e., have had bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least six months prior to first dose of PRX-00023; appropriate documentation will be required) OR (b) Agree that, if sexually active, they and all male partners will use two (2) acceptable barrier forms of contraception (e.g., condoms and diaphragm) from screening until one month after the final dose of study drug
* Male subjects must agree that they and any female partners will use two(2) acceptable forms of contraception (e.g., condoms and hormonal contraceptives) from screening until one month following the final dose of study drug
* Be in generally good physical health as determined by the Investigator on the basis of medical history, physical examination, and screening laboratory results
* Have the ability to communicate with the investigative site staff in a manner sufficient to carry out all protocol procedures as described
* Be able to understand procedures and provide written informed consent prior to admission

Exclusion Criteria:

* A history of an inability to tolerate, or a failure to respond to, two or more anxiolytic or anti-depressant drugs given in adequate doses and duration for the treatment of symptoms present in the current illness
* Prior intolerance to buspirone, gepirone, tandospirone or other 5HT1A agonist
* A current or past history of mania, bipolar disorder, schizophrenia, or other psychotic disorder
* A current history (or within the six months prior to screening) of panic disorder, post traumatic stress disorder, major depression, obsessive-compulsive disorder, social phobia, acute stress disorder, adjustment disorder with anxious mood, performance anxiety, somatization disorder, or other principle psychiatric diagnosis (DSM-IV) which could interfere with the efficacy assessments
* A history of a major life event (e.g. divorce, death of family member) which in the opinion of the Investigator is likely to alter the efficacy ratings during the course of the study
* Clinically significant abnormalities on laboratory tests or ECG (includes QTc value >450 msec in males or > 470 msec in females)
* The presence of a serious or clinically unstable neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematologic or other medical illness or psychiatric condition that would, in the opinion of the Investigator, compromise participation in the study, confound study results, or likely lead to the need for early termination of study participation or hospitalization during the course of the study
* A history of allergic reactions to two or more medications of different chemical classes
* Use of any non-prescription drug with psychotropic effects within seven (7) days prior to initiation of the placebo lead in
* Chronic use of analgesics with opiates (e.g., codeine, hydrocodone, oxycodone) for >6 months or use of opiates within two weeks prior to screening
* Introduction or change in cognitive behavioral therapy, interpersonal therapy, or other psychotherapy within three months of screening
* Use of St. John's Wort, kava kava, ephedra, or other psychoactive herbal medications within the last two weeks before screening
* Known or suspected substance abuse or dependence, including alcohol, within one year of screening
* A positive urine drug screen (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, methaqualone, opiates, and propoxyphene) at screening. The urine drug screen may be repeated once if after discussion with the patient there is a plausible reason for the positive test other than substance abuse
* A history of suicide attempts in the last two years, or current suicide risk in the judgment of the Investigator
* Women who are breast feeding, have been lactating within three months prior to screening, pregnant, expect to become pregnant during the course of the study, or are sexually active and are not using a medically acceptable double barrier method of birth control. Women relying solely on oral contraceptives for - The use of any investigational drug within 30 days prior to enrollment
* The concomitant use of any other antidepressants, anxiolytics, or any other psychoactive drugs
* Treatment with any potent inhibitor of CYP3A4, including ketoconazole, itraconazole, HIV protease inhibitors, clarithromycin, erythromycin, cyclosporine
* Treatment with CYP3A4 inducers such as carbamazepine, barbiturates, phenytoin, rifampin, or oral glucocorticoids
* Treatment with any of the psychoactive drugs listed in the table below within the interval specified below before enrollment
* Psychoactive drug - Interval (weeks)

  * MAO Inhibitors - 4
  * Fluoxetine - 4
  * Fluvoxamine - 2
  * Citalopram - 2
  * Paroxetine - 2
  * Sertraline - 2
  * Buspirone - 4
  * Buproprion - 2
  * Mirtazepine - 2
  * Nefazodone - 2
  * Venlafaxine - 2
  * Duloxetine - 2
  * Trazodone - 2
  * Benzodiazepines Occasional or PRN use: - 1
  * Chronic or daily use: - 4
  * Tricyclic and Heterocyclic Antidepressants - 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310
Dates: Start 2005-08; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Vista Medical Research, Mesa, Arizona
  - Pivotal Research Center, Mesa, Arizona
  - Anaheim Research Center, Anaheim, California
  - Pacific Clinical Research Group, Upland, California
  - Connecticut Clinical Research, Cromwell, Connecticut
  - The George Washington University, Washington D.C., District of Columbia
  - Gulf Coast Clinical Research Center, Fort Myers, Florida
  - Atlanta Institute of Research and Medicine, Atlanta, Georgia
  - Northwest Behavioral Research, Marietta, Georgia
  - Louisiana Research Associates, New Orleans, Louisiana
  - Pivotal Research Center, Royal Oak, Michigan
  - Comprehensive Neurosciences, Kenilworth, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Oregon Center for Clinical Investigations, Portland, Oregon
  - Oregon Center for Clinical Investigations, Salem, Oregon
  - Unversity of Pennsylvania, Philadelphia, Pennsylvania
  - Future Search Trials, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Comprehensive Neurosciences, Falls Church, Virginia
  - Sidney Lerfald, MD, Charleston, West Virginia